CLINICAL TRIAL: NCT04647552
Title: The Effect of Hydrocortison Treatment on Angiotensin II and Angiotensin Receptors in Patients Suffering From Septic Shock: A Prospective Observational Study
Brief Title: Effects of Hydrocortison Treatment on Angiotensin II and Angiotensin II Receptors in Patients With Septic Shock
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ayse Belin Ozer, Prof. Dr., Inonu University
Other Study IDs: AOzer
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Shock, Septic
Keywords: Shock, Septic; hydrocortisone; angiotensin II
MeSH Terms: conditions — Shock, Septic | interventions — Hydrocortisone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- hydrocortisone: The patients with septic shock who required a noradrenaline infusion rate above 0.5µg/kg
  Interventions: Drug: Drug Steroid
- control: The patients with septic shock who needed a noradrenaline infusion rate of up to 0.5µg/kg/min to maintain MAP>65 mmHg

INTERVENTIONS:
Drug: Drug Steroid — hydrocortisone injection
  Other Names: hydrocortisone
  Groups: hydrocortisone

SUMMARY:
This study aims to evaluate the role of angiotensin II, AT1, and AT2 on catecholomine responsive and catecholomine resistant septic shock, and the effect of hydrocortisone traetment on catecholomine resistant septic shock and angiotensin II, AT1, and AT2.Angiotensin II can be used as a biomarker of vasoplegia observed in refractory septic shock unresponsive to catecholamine. In these patients; therapeutic effect of hydrocortisone on hypotension was performed by decreasing AT 2 level, AT2 should be investigated as a therapeutic target in the treatment of vasoplegia-induced hypotension and SVRI measured by minimally invasive cardiac output method suggests that it can be used as a useful parameter in the diagnosis and follow-up of vasoplegia.

DETAILED DESCRIPTION:
This study will be enrolled 40 patients diagnosed with septic shock according to Sepsis 3 criteria. The patients with septic shock who needed a noradrenaline infusion rate of up to 0.5µg/kg/min to maintain MAP>65 mmHg will be classified as control group (n=20) and the ones who required a noradrenaline infusion rate above 0.5µg/kg will be classified as hydrocortisone group (n=20). Blood samples will be taken for analysis of plasma angiotensin II, AT1, AT2 levels at the time of diagnosis, one hour after and on the 3rd day of the bundle and the hydrocortisone treatment. Hemodynamic parameters simultaneously obtain by continuous minimal invasive cardiac output measurement method will record.

ELIGIBILITY:
Inclusion Criteria:

* septic shock patient

Exclusion Criteria:

* other causes of end-stage organ failure, immunodeficiency, presence of acute mesenteric ischemia, vasospastic disease, pregnancy, other shock causes (hypovolemic, cardiogenic, neurogenic), life expectancy less than 48 hours corticosteroid use in the last 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was enrolled 40 patients diagnosed with septic shock according to Sepsis 3 criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Serum angiotensin II levels | 0-3 days
  Serum angiotensin II levels
Serum angiotensin II reseptor 1 levels | 0-3 days
  Serum angiotensin II reseptor 1 levels
Serum angiotensin II reseptor 2 levels | 0-3 days
  Serum angiotensin II reseptor 2 levels

SECONDARY OUTCOMES:
Mortality rate | 28 days
  mortality rate
SVRI | 0-3 days
  systemic vascular resistans index

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Belin B OZER, Principal Investigator — Inonu University Faculty of Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Ayse Belin B OZER, Malatya
  - Ayse Belin OZER, Malatya

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Zhang W, Chen X, Huang L, Lu N, Zhou L, Wu G, Chen Y. Severe sepsis: Low expression of the renin-angiotensin system is associated with poor prognosis. Exp Ther Med. 2014 May;7(5):1342-1348. doi: 10.3892/etm.2014.1566. Epub 2014 Feb 20. PMID 24940436